CLINICAL TRIAL: NCT01608048
Title: Transcutaneous Electrical Acupoint Stimulation to Improve Pregnancy Rates for Women Undergoing in Vitro Fertilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Cui Hong Zheng, assistant research fellow, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZheng2012QN180
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2012-11

CONDITIONS: Supervision of Pregnancy Resulting From In-vitro Fertilization
Keywords: In-vitro Fertilization; transcutaneous electrical acupoint stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention)
- TEAS (Experimental)
  Interventions: Device: transcutaneous electrical acupoint stimulation (TEAS);EA
- EA:electro-acupuncture (Experimental)
  Interventions: Device: transcutaneous electrical acupoint stimulation (TEAS);EA

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation (TEAS);EA — TEAS group (conventional IVF + TEAS), electro-acupuncture (EA) group (conventional IVF + electro-Acu.), and control group (only conventional IVF) Parameter of TEAS or EA: frequency of 2/100 Hz；moderate electrical current. Treatments start from the day 3 of menstruation，once every two days, 30 min for each for two continuous weeks.
  Arms: EA:electro-acupuncture; TEAS

SUMMARY:
The objective of this study is to investigate the effect of transcutaneous electrical acupoint stimulation on pregnancy rates in women undergoing in vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

(1) infertile women < 40 years of age, undergoing a fresh IVF or intracytoplasmic sperm injection (ICSI) cycle; (2) be an appropriate candidate with the potential for a lower success rate which defined as two or more previous unsuccessful ETs (fresh or frozen); (3) are willing to sign an informed consent form, indicating that they are aware of the investigational nature of this study that is in keeping with the policies of the institution; (4) willing to return to the study site for their study visits. The reason for our inclusion criteria is that women experienced several unsuccessful OAs or ETs may easily accept randomization to this study, and for whom adding TEAS or EA may significantly improve their clinical outcomes.

Exclusion Criteria:

(1) major medical illnesses (like stage III heart disease, severe hypertension, uncontrolled diabetes mellitus, HIV positivity, severe bleeding dyscrasias, etc.) possibly precluding IVF or pregnancy; (2) FSH more than 20 IU/L; (3) receiving donor eggs; (4) cutaneous lesion of certain acupoint area; (5) having been previously participated in this study or having undertaken acupuncture (in whatever modality) treatment for infertility.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate (CPR) | 1 year

SECONDARY OUTCOMES:
Live birth rate (LBR) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cui Hong Zheng, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- IVF center of Tongji Hospital,Tongji medical college,HUST, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zheng CH, Zhang J, Wu J, Zhang MM. The effect of transcutaneous electrical acupoint stimulation on pregnancy rates in women undergoing in vitro fertilization: a study protocol for a randomized controlled trial. Trials. 2014 May 9;15:162. doi: 10.1186/1745-6215-15-162. PMID 24886647